CLINICAL TRIAL: NCT00428337
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of DNA Vaccine EP-1233 and Recombinant MVA-HIV Polytope Vaccine MVA-mBN32, Separately and in a Combined Prime-boost Regimen, When Given to Healthy, Vaccinia-naive, HIV-1-uninfected Adults
Brief Title: Safety of and Immune Response to a DNA Vaccine and a Recombinant HIV-1-MVA Vaccine, Separately and in Combination, in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); Pharmexa-Epimmune (Unknown); Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 067; 10394 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; EP1233; MVA-mBN32; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Participants will receive one injection of DNA vaccine EP-1233 or placebo in each shoulder on Days 0 and 28 and one injection of MVA-mBN32 or placebo in each arm on Days 84 and 168
  Interventions: Biological: EP-1233; Biological: MVA-mBN32
- 2 (Experimental): Participants will receive one injection of DNA vaccine EP-1233 or placebo in each shoulder on Days 0, 28, 84, and 168
  Interventions: Biological: EP-1233
- 3 (Experimental): Participants will receive one injection of MVA-mBN32 or placebo in each arm on Days 0, 28, 84, and 168
  Interventions: Biological: MVA-mBN32

INTERVENTIONS:
Biological: EP-1233 — DNA-HIV-recombinant vaccine
  Arms: 1; 2
Biological: MVA-mBN32 — HIV-recombinant viral vaccine
  Arms: 1; 3

SUMMARY:
The purpose of this study is to determine the safety of and immune response to two experimental vaccines, designed for use in combination, for the prevention of HIV infection in healthy adults.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through the development of a safe and effective vaccine that will prevent HIV infection. DNA-based vaccines alone promote a weak immune response but when used as priming immunogens, followed by a recombinant viral vaccine that is a very attenuated vaccinia (smallpox) vaccine presenting the same immunogens as a booster, immunization with such a combination regimen seems to induce much stronger responses. EP-1233 is a DNA-HIV-recombinant vaccine designed to interact with CD4 (helper-inducer) and CD8 (cytotoxic) T lymphocytes (T cells) to prime CD4 and CD8 cells to respond to HIV components. MVA-mBN32 is a HIV-recombinant viral (MVA) vaccine that through other ways of interacting with CD4 and CD8 cells to immunize (boost) with similar HIV immunogens, may result in a stronger immune response.

The purpose of this study is to determine the safety of and immune response to two experimental vaccines for the prevention of HIV infection, individually and in combination, in healthy adults who have not been previously vaccinated against smallpox. Participants will be randomly assigned to one of three groups. All participants will receive injections at Days 0, 28, 84, and 168 of the study. Participants assigned to Group 1 will receive, on Day 0, one injection in each arm of EP-1233 or placebo and the same study product (EP-1233 or the DNA placebo) on Day 28. Thereafter, each Group 1 participant will receive one injection of MVA-mBN32 or placebo on Days 84 and 168. Groups 2 and 3 will not begin enrollment until safety and immunogenicity data from Group 1 have been evaluated. Participants assigned to Group 2 will receive only the DNA vaccine EP-1233 (or placebo) in each arm on all injection days. Participants in Group 3 will not begin enrollment until safety and immunogenicity data from Group 1 have been evaluated. Participants assigned to Group 3 will receive a consistent regimen of MVA-mBN32 (or placebo) on all injection days. Participants will be required to keep a symptom log for 3 days after each injection and attend clinical visits on Day 0, 14, 28, 42, 84, 98, 168, 182, 273, and 364 of the study. At each of the 10 visits, a physical exam, cardiac assessment, and HIV risk reduction and prevention counseling will occur. Blood collection will occur on Days 0, 14, 42, 98, 182, 273, and 364. Urine collection will occur on Days 14, 42, 98, and 182.

ELIGIBILITY:
Inclusion Criteria:

* Good general health

Exclusion Criteria:

* Previous receipt of smallpox vaccination
* HIV-infected
* Hepatitis B surface antigen positive
* Participation in prior HIV vaccination trial
* Immunosuppressive medications within 168 days prior to study entry
* Receipt of blood products within 120 days of study entry
* Receipt of live attenuated, medically indicated subunit, or killed (inactivated) vaccines within 30 days of study entry
* Certain abnormal lab values
* Pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-04; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety of vaccination, as measured by number of adverse events, local and systemic reactogenicity signs and symptoms, changes in electrocardiogram (ECG), cardiac troponin I levels, and differences in other safety laboratory measures | Throughout study

SECONDARY OUTCOMES:
HIV-specific intracellular cytokine staining (ICS) assay and/or interferon-gamma ELISA responses | At 2 weeks following the third and fourth injection
Vaccinia-specific neutralizing binding assays performed on serum samples from participants receiving the MVA vaccine | At 2 weeks following the final vaccination
Self reports on social impact of participation in study | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Gorse, Study Chair — Saint Louis University School of Medicine; Christine Mhorag Hay, Study Chair — University of Rochester
Locations (3):
- United States (3):
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - Vanderbilt Vaccine CRS, Nashville, Tennessee

REFERENCES:
- [Background] Dale CJ, Thomson S, De Rose R, Ranasinghe C, Medveczky CJ, Pamungkas J, Boyle DB, Ramshaw IA, Kent SJ. Prime-boost strategies in DNA vaccines. Methods Mol Med. 2006;127:171-97. doi: 10.1385/1-59745-168-1:171. PMID 16988455
- [Background] Ostrowski MA, Yu Q, Yue FY, Liu J, Jones B, Gu XX, Loutfy M, Kovacs CM, Halpenny R. Why can't the immune system control HIV-1? Defining HIV-1-specific CD4+ T cell immunity in order to develop strategies to enhance viral immunity. Immunol Res. 2006;35(1-2):89-102. doi: 10.1385/IR:35:1:89. PMID 17003512
- [Background] Rodriguez-Chavez IR, Allen M, Hill EL, Sheets RL, Pensiero M, Bradac JA, D'Souza MP. Current advances and challenges in HIV-1 vaccines. Curr HIV/AIDS Rep. 2006 Feb;3(1):39-47. doi: 10.1007/s11904-006-0007-0. PMID 16522258
- [Derived] Elizaga ML, Vasan S, Marovich MA, Sato AH, Lawrence DN, Chaitman BR, Frey SE, Keefer MC; MVA Cardiac Safety Working Group. Prospective surveillance for cardiac adverse events in healthy adults receiving modified vaccinia Ankara vaccines: a systematic review. PLoS One. 2013;8(1):e54407. doi: 10.1371/journal.pone.0054407. Epub 2013 Jan 17. PMID 23349878